CLINICAL TRIAL: NCT01603446
Title: Pilot Study to Investigate the Efficacy of L-arginine Therapy on Endothelium-dependent Vasodilation & Mitochondrial Metabolism in MELAS Syndrome.
Brief Title: L-arginine Therapy on Endothelium-dependent Vasodilation & Mitochondrial Metabolism in MELAS Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Ingrid Tein, Staff Neurologist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000023405
Record Dates: First submitted 2012-05-18; First posted 2012-05-22 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: MELAS Syndrome
Keywords: pediatric; MELAS; mechanism of action of L-arginine
MeSH Terms: conditions — MELAS Syndrome | interventions — Arginine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MELAS Patients (Experimental): Three siblings with MELAS (A3243G) syndrome (1 male; 2 females) aged 17-23 years, followed or previously followed in the Neurometabolic Clinic at the Hospital for Sick Children will be studied.
  Interventions: Drug: L-Arginine
- Control Group (No Intervention): Four age- and sex-matched controls and female controls will be matched according to phase in menstrual cycle corresponding with their age-matched MELAS subjects

INTERVENTIONS:
Drug: L-Arginine — NOW® L-Arginine powder
  Arms: MELAS Patients

SUMMARY:
MELAS patients suffer from exercise intolerance, weakness, poor vision or blindness, poor growth, developmental delay, and deafness. They also have unique 'stroke-like' episodes (SLEs) which are not due to blockages of large or medium arteries. These 'strokes' are thought to be due to energy failure of very small brain blood vessels combined with energy failure in the mitochondria (cell battery) of the brain cells, especially in the back region of the brain in the vision centre. This leads to visual loss and paralysis. The overall goal of this study is to better understand the mechanism of these SLEs at the level of the brain cells and small blood vessels.

DETAILED DESCRIPTION:
We will study a family of 3 siblings, each with different severities of MELAS, using safe, non-invasive tests. We will determine whether there is a decrease in the ability of small brain blood vessels to increase blood flow by dilating in response to certain stimuli such as increased blood carbon dioxide levels or in response to brain cell activation in the vision centre by visual stimuli. We will use a technique called BOLD-fMRI which can detect changes in brain blood flow. As exercising muscle also depends on increased blood flow and mitochondrial energy, we will study different measures of aerobic energy metabolism in exercising muscle using cycle exercise testing and special phosphorus-magnetic resonance spectroscopy which measures the changes in the major chemicals of muscle energy metabolism. The dietary amino acid L-arginine is known to dilate blood vessels increasing blood flow and to decrease toxic free radicals that are generated by dysfunctional mitochondria. We will determine the effect of a single dose and a 6 week trial of oral L-arginine, on brain blood vessel reactivity, brain cell activation and muscle aerobic function to see how useful this would be in the treatment of these patients and other mitochondrial disorders which present with strokes.

ELIGIBILITY:
Inclusion Criteria:

Experimental Siblings with MELAS (A3243G) syndrome

* 17-23 years
* Followed Neurometabolic Clinic at the Hospital for Sick Children will be studied.
* Normal electrolytes, glucose, renal and liver functions & no history of gastrointestinal, respiratory or cardiac problems.

Controls

-Aged 17-23- Sex matched to the MELAS subjects

Exclusion Criteria:

Controls

* Experience migraines
* Have a metabolic disorder
* Taking medications predisposing to lactic acidosis or vasodilatation
* Neuromuscular/neurologic condition
* Cardiac or pulmonary disease
* Visual abnormalities
* Hypertension, anemia and prothrombotic state. Control subjects
* Contraindication for MRI (pacemaker, ocular metal, claustrophobia, tattoos) will be excluded from the study.

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Muscle function investigation via 31P-Magnetic resonance spectroscopy | 60 to 105 minutes post dose
  We will study exercising quadriceps using our MR-compatible up-down ergometer and our well established aerobic exercise protocol at 65 % of maximal voluntary contraction.

SECONDARY OUTCOMES:
Total body maximal aerobic capacity | 60-75 mins post dose
  Maximal incremental cycle ergometry is conducted in our CardioRespiratory Exercise Lab at HSC by our established protocols (26). Serum CK and quantitative AA (for arginine, ornithine and citrulline) will be measured pre- and post- exercise as well as eNO in order to correlate aerobic exercise parameters with serum arg and eNO levels..
CerebroVascular Reactivity | 75-105 mins post dose
  Functional MRI-Blood oxygen level dependent (BOLD) of brain
Exhaled Nitric Oxide (eNO) | 75 mins pre dose, 75 mins post dose
  eNO will be measured using single breath on-line measurements for the assessment of lower airway Nitric Oxide

CONTACTS AND LOCATIONS:
Overall Officials: Ingrid Tein, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Rodan LH, Poublanc J, Fisher JA, Sobczyk O, Mikulis DJ, Tein I. L-arginine effects on cerebrovascular reactivity, perfusion and neurovascular coupling in MELAS (mitochondrial encephalomyopathy with lactic acidosis and stroke-like episodes) syndrome. PLoS One. 2020 Sep 3;15(9):e0238224. doi: 10.1371/journal.pone.0238224. eCollection 2020. PMID 32881886
- [Derived] Rodan LH, Wells GD, Banks L, Thompson S, Schneiderman JE, Tein I. L-Arginine Affects Aerobic Capacity and Muscle Metabolism in MELAS (Mitochondrial Encephalomyopathy, Lactic Acidosis and Stroke-Like Episodes) Syndrome. PLoS One. 2015 May 20;10(5):e0127066. doi: 10.1371/journal.pone.0127066. eCollection 2015. PMID 25993630